CLINICAL TRIAL: NCT02207127
Title: Magnetic Resonance Imaging in Obstructive Sleep Apnea
Acronym: MRI in OSA
Status: Withdrawn | Type: Observational
Why Stopped: Unable to refine study measurements/protocol adequately.
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HS-14-00101
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI, DISE, and Surgery: All participants will undergo MRI and DISE prior to undergoing surgical treatment of obstructive sleep apnea.
  Interventions: Procedure: MRI, DISE, and Surgery

INTERVENTIONS:
Procedure: MRI, DISE, and Surgery — MRI, DISE, and Surgery

SUMMARY:
There is a fundamental gap in the investigators ability to design effective surgical treatment of obstructive sleep apnea (OSA) for the 30-40% of patients who cannot tolerate non-surgical treatment. OSA surgery outcomes vary widely, with the chances of a successful outcome ranging from 5% to 65% for individual or combination procedures. To predict - and thereby to improve - outcomes, the investigators must determine what predicts surgical success. This project will compare findings from two evaluations: drug-induced sleep endoscopy (DISE) and upper airway magnetic resonance imaging (MRI). DISE has demonstrated important benefits, but it has important limitations. Upper airway MRI is the most complete evaluation performed during wakefulness, making it conducive to broad application and less expensive than DISE, but there are no studies utilizing MRI as a surgical evaluation. The investigators propose a cross-sectional analysis of 40 adult subjects with moderate to severe OSA. In addition to history, physical examination, and polysomnogram (sleep study), all subjects will undergo DISE and MRI to characterize the pattern of obstruction. The investigators will examine the association between DISE and MRI, focusing on specific DISE findings that have been associated with surgical outcomes. The investigators multidisciplinary team has substantial expertise and experience in OSA investigation, DISE, and upper airway MRI.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 21 years; moderate to severe OSA (AHI ≥15 events/hour)
* body mass index <40 kg/m2.

Exclusion Criteria:

* prior OSA surgery
* known neurologic, cardiac, pulmonary, renal, or hepatic disorders
* psychiatric problems except for treated depression or mild anxiety
* co-existing sleep disorder other than OSA
* other contraindication to DISE or MRI such as propofol allergy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be adults with obstructive sleep apnea undergoing surgery. All participants will undergo magnetic resonance imaging (MRI) and drug-induced sleep endoscopy (DISE).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Surgical results | 6 months
  Surgical outcomes will be measured using sleep study outcomes (apnea-hypopnea index). The analysis will include evaluation of a potential association between surgical outcomes and both MRI and DISE measures.

SECONDARY OUTCOMES:
Sleep-Related Quality of Life | 6 months
  Sleep-related quality of life will be assessed with the Functional Outcomes of Sleep Questionnaire. Changes will be determined by a comparison of preoperative and postoperative scores.
Daytime Sleepiness | 6 months
  Daytime sleepiness will be assessed with the Epworth Sleepiness Scale score. Changes will be determined by a comparison of preoperative and postoperative scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Hospital of USC, Los Angeles, California, United States